CLINICAL TRIAL: NCT02734329
Title: Zero Ischemia Laparoscopic Radio Frequency/Microwave Ablation Assisted Enucleation of Renal Cell Carcinoma With T1 Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Changzheng Hospital (Other); Changhai Hospital (Other); Shanghai 6th People's Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Yiran Huang, Director of Urology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-2016006
Record Dates: First submitted 2016-02-29; First posted 2016-04-12 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Neoplasms
Keywords: Nephron sparing surgery; Zero ischemia; Warm ischemia; Laparoscopic; Radiofrequency ablation; Microwave ablation
MeSH Terms: conditions — Kidney Neoplasms

ARMS (2):
- Zero Ischemia group (Experimental): Radiofrequency ablation(RFA) /Microwave ablation(MVA) will be performed for 1 to 4 cycles each depending on tumor size and depth. The tumor then will be laparoscopic enucleation without hilar clamping in most cases.
  Interventions: Procedure: zero ischemia laparoscopic RFA/MVA assisted tumor enucleation (TE)
- Conventional group (Active Comparator): Renal hilum will be accurately isolated and then the artery only will be clamped during surgery.
  Interventions: Procedure: conventional laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: conventional laparoscopic partial nephrectomy — renal artery will be clamped during surgery.
  Arms: Conventional group
Procedure: zero ischemia laparoscopic RFA/MVA assisted tumor enucleation (TE)
  Arms: Zero Ischemia group

SUMMARY:
Zero ischemia laparoscopic radio frequency ablation assisted tumor enucleation has been proved to enable tumor excision with relatively better renal function preservation comparing with conventional laparoscopic partial nephrectomy for T1a renal cell carcinoma (RCC) in a randomized clinical trial in single center. The investigators want to explore this technique to T1 RCC patients in randomized clinical trial in multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* patients with sporadic, unilateral, newly diagnosed T1 presumed renal cell carcinoma
* patients scheduled for laparoscopic nephron sparing surgery
* patients agreeable to participate in this long-term follow-up study

Exclusion Criteria:

* patients' aged >80 years
* patients with other renal diseases,(including kidney stone, glomerular nephritis, etc.) which might affect the renal function of the operative kidney
* patients not able to tolerate the laparoscopic procedure
* patients with previous renal surgery or history of any inﬂammatory conditions of the operative kidney
* patients with the renal tumor involving urinary collecting system

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the change in glomerular ﬁltration rate (GFR) of the affected kidney | Baseline and 30 months
changes of estimated GFR (eGFR) | Baseline and 30 months

SECONDARY OUTCOMES:
estimated blood loss | during surgery
rates of positive surgical margin | postoperative，up to 2 weeks after surgery
postoperative complications | postoperative，up to 30 days
the rate of local recurrence | through study completion, an average of 3 years
operative time | During surgery
Hospital stay time | The time from the surgery day to patient discharge, up to 2 weeks
progression-free survival rate | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China